CLINICAL TRIAL: NCT06313112
Title: Utilization of Maternal Health Services, Birth Outcomes and Infant Growth and Its Linkage With Food Insecurity Among Slum-Dwelling Women in Pune, India
Brief Title: Impact of Food Insecurity on Utilization of Maternal Healthcare Services and Birth Outcomes in Slums in Pune, India
Acronym: MCH
Status: Active, not recruiting | Type: Observational
Sponsor: Hirabai Cowasji Jehangir Medical Research Institute (Other)
Responsible Party: Principal Investigator, Dr. Anuradha Khadilkar, Deputy Directors, Hirabai Cowasji Jehangir Medical Research Institute
Other Study IDs: JCDC/BHR/23/036
Record Dates: First submitted 2024-02-23; First posted 2024-03-15 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Prenatal Care; Food Insecurity; Pregnancy Outcome
Keywords: Prenatal Care; Antenatal Care; Healthcare; Postnatal Care; Household Food Insecurity; Birth Outcomes
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational study — Observational study

SUMMARY:
The goal of this observational study is to assess household food insecurity among slum-dwelling women in India and to explore if household food insecurity is associated with utilization of maternal healthcare services, birth outcomes and infant growth.

The main questions it aims to answer are:

* Is the utilization of maternal healthcare services antenatally, during delivery, and postnatally associated with household food insecurity among slum-dwelling women in Pune, India?
* Is household food insecurity associated with birth outcomes and infant growth in these women?

Participants will be asked:

* For information related to socio-demographic characteristics, healthcare services utilization, food insecurity experience, dietary intake, and infant feeding indicators using a questionnaire.
* Anthropometric measurements of the participant, her husband and her infant/s will be collected.
* Two focused group discussions (FGDs) will also be conducted to gain insight into the perceptions of these women with respect to the utilization of maternal healthcare services. One FGD will be conducted for women who availed all the healthcare services and the other for those who did not adequately avail of the antenatal and postnatal services.

DETAILED DESCRIPTION:
The first target indicator of Sustainable Development Goals (SDG) 3 i.e Good Health and Well-being for all at all ages is reducing the global maternal mortality ratio (MMR) to less than 70 per 100,000 live births by 2030. While there had been a significant reduction in the MMR globally from 385 maternal deaths per 100,000 live births in 1990 to 211 maternal deaths per 100,000 live births in 2017, the MMR increased slightly to 223 deaths per 100,000 live births in 2020. India, however, has been performing well on this indicator with progressive reduction in MMR from 130 deaths per 100,000 live births in 2014-16 to 97 deaths per 100,000 live births in 2018-2020, with eight Indian states achieving the SDG target of MMR < 70. Maharashtra ranks 2nd among these eight states with an MMR of 33 in 2018-2020. In spite of the stellar progress made by India, together with Nigeria it still accounted for one-third of the global MMR contributing to 8% of the total maternal deaths in 2020, and India also accounted for nearly two-thirds of the MMR in the South East Asia region.

It is well-known that the appropriate utilization of maternal healthcare services contributes to reduced maternal morbidity and mortality and improved offspring health. It has also been established that utilization of one of the services in the continuum of care for maternal and child health greatly increases the likelihood of utilization of the subsequent services. For example, women who availed of even one ANC visit were more likely to opt for institutional deliveries and postnatal care. India provides comprehensive continuum of care in maternal and newborn health comprising quality antenatal care (ANC), delivery care, and postnatal care (PNC). However, there is considerable regional inequity in the utilization of these services. There are multiple factors that influence the utilization of maternal healthcare services which vary by region, religion, socio-economic status, and service delivery environment among many others. Thus, it is imperative to identify enablers, barriers and need gaps location wise so that appropriate interventions can be developed for promotion of healthcare service utilization.

Considering the rapid proliferation of the slum population in India, and also Pune, household food insecurity is proving to be a major challenge due to competition among the informal workforce residing in slums for basic life necessities. In particular, food insecurity negatively impacts pregnant and lactating women as gender biases may interfere with their access to adequate food thus, affecting their health and the health of their offspring. Food insecurity may cause people to prioritize activities that enable them to gain access to food over health seeking. This may result in poor utilization of maternal healthcare services which may be difficult to access or may involve costs and time in accessing them. Thus, the investigators deemed it necessary to assess household food insecurity among slum-dwelling women in India and to explore if household food insecurity is associated with maternal healthcare services utilization.

The objectives of the study are as follows:

1. To assess the utilization of antenatal and postnatal health care services by slum-dwelling women from Pune
2. To explore the association of utilization of maternal healthcare services ante and postnatally with birth outcomes and infant growth
3. To examine the association of household food insecurity with maternal healthcare service utilization, birth outcomes and infant growth

ELIGIBILITY:
Inclusion Criteria:

A woman will be recruited in the study if she

1. is willing and able to give an informed consent
2. has been residing in a slum for a minimum of 2 years
3. is aged between 18 to 49 years
4. has an infant or infants between 1.5 to 6 months of age

Exclusion Criteria:

A subject will not be eligible for inclusion in this study if any of the following criteria apply:

1. She is unwilling to consent to participate in the study
2. The age of her infant is less than 1.5 months or greater than 6 months.
3. Her infant has any congenital conditions

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Slum dwelling women who have infants aged 1.5 months to 6 months
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2023-10-09 (Actual); Primary Completion 2024-07-16 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of women who availed at least three Antenatal Care (ANC) visits | Through study completion, an average of 1 year
  Percentage of women who availed at least three Antenatal Care (ANC) visits
Percentage of women who had contact with Accredited Social Health Activist (ASHA) worker during pregnancy | Through study completion, an average of 1 year
  Percentage of women who had contact with ASHA worker during pregnancy
Percentage of women who consumed at least 100 Iron Folic Acid tablets | Through study completion, an average of 1 year
  Percentage of women who consumed at least 100 Iron Folic Acid tablets
Percentage of women who consumed deworming tablets at least once during pregnancy | Through study completion, an average of 1 year
  Percentage of women who consumed deworming tablets at least once during pregnancy
Percentage of women who underwent delivery preparedness | Through study completion, an average of 1 year
  Percentage of women who underwent delivery preparedness
Percentage of women with knowledge of key danger signs during pregnancy | Through study completion, an average of 1 year
  Percentage of women with knowledge of key danger signs during pregnancy such as vaginal bleeding, severe headaches
Percentage of women who delivered at institution | Through study completion, an average of 1 year
  Percentage of women who delivered at institution
Percentage of women who stayed at a facility for at least 24 hours post-delivery | Through study completion, an average of 1 year
  Percentage of women who stayed at a facility for at least 24 hours post-delivery
Percentage of women who received post-natal care within a week of delivery | Through study completion, an average of 1 year
  Percentage of women who received post-natal care within a week of delivery

SECONDARY OUTCOMES:
Association of demographic characteristics and household food insecurity scores with the indicators of utilization of healthcare services | Through study completion, an average of 1 year
  The association of demographic characteristics such as age of the participant, education of participant and her husband, occupation of participant and her husband, socio-economic status of the family, gender of the infant and household food insecurity scores will be investigated with each indicator of utilization of maternal healthcare service.

OTHER OUTCOMES:
Correlation of indicators of utilization of healthcare services with birth outcomes | Through study completion, an average of 1 year
  Correlation of the indicators of utilization of healthcare services with birth outcomes such as
  1. gestational age at birth - preterm or term birth
  2. birth weight - low birth weight or appropriate birth weight
  3. gestational size - small for gestational age / appropriate for gestational age
  4. Neonatal complications
Correlation of indicators of utilization of healthcare services with infant growth | Through study completion, an average of 1 year
  Correlation of the indicators of utilization of healthcare services with infant growth parameters such as
  1. body weight
  2. length
  3. mid-upper arm circumference

CONTACTS AND LOCATIONS:
Overall Officials: Rubina M Mandlik, PhD, Principal Investigator — Hirabai Cowasji Jehangir Medical Research Institute Pune
Locations (1):
- Hirabai Cowasji Jehangir Medical Research Institute, Pune, Maharashtra, India

IPD SHARING:
Plan to Share IPD: Undecided